CLINICAL TRIAL: NCT02605174
Title: A Study of Three Doses of Lasmiditan (50 mg, 100 mg and 200 mg) Compared to Placebo in the Acute TReaTment of MigrAiNe: A Randomized, Double-blind, Placebo-controlled Parallel Group Study (SPARTAN)
Brief Title: Three Doses of Lasmiditan (50 mg, 100 mg and 200 mg) Compared to Placebo in the Acute Treatment of Migraine
Acronym: SPARTAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: CoLucid Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 16889; H8H-CD-LAHK (Other: Eli Lilly and Company); 2015-005689-40 (EudraCT Number); COL MIG-302 (Other: Colucid)
Record Dates: First submitted 2015-11-11; First posted 2015-11-16 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Migraine With or Without Aura
MeSH Terms: interventions — lasmiditan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lasmiditan 50 milligram (mg) (Experimental): Oral tablet. Lasmiditan 50 mg plus placebo (to match a lasmiditan dose). One dose for acute treatment of migraine. Second dose for rescue or recurrence of migraine allowed between 2 and 24 hours.
  Interventions: Drug: Lasmiditan 50 mg
- Lasmiditan 100 mg (Experimental): Oral tablet. Lasmiditan 100 mg plus placebo (to match a lasmiditan dose). One dose for acute treatment of migraine. Second dose for rescue or recurrence of migraine allowed between 2 and 24 hours.
  Interventions: Drug: Lasmiditan 100 mg
- Lasmiditan 200 mg (Experimental): Oral tablet. Lasmiditan 200 mg plus placebo (to match a lasmiditan dose). One dose for acute treatment of migraine. Second dose for rescue or recurrence of migraine allowed between 2 and 24 hours.
  Interventions: Drug: Lasmiditan 200 mg
- Placebo (Placebo Comparator): Oral tablet. Placebo tablets match each of the lasmiditan doses (50 mg, 100 mg and 200 mg). One dose for acute treatment of migraine. Second dose for rescue or recurrence of migraine allowed between 2 and 24 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lasmiditan 50 mg — One tablet lasmiditan 50 mg plus one placebo tablet (matching one of the lasmiditan doses)
  Other Names: LY573144
  Arms: Lasmiditan 50 milligram (mg)
Drug: Lasmiditan 100 mg — One tablet lasmiditan 100 mg plus one placebo tablet (matching one of the lasmiditan doses)
  Other Names: LY573144
  Arms: Lasmiditan 100 mg
Drug: Lasmiditan 200 mg — One tablet lasmiditan 200 mg plus one placebo tablet (matching one of the lasmiditan doses)
  Other Names: LY573144
  Arms: Lasmiditan 200 mg
Drug: Placebo — Two placebo tablets to match lasmiditan doses.
  Arms: Placebo

SUMMARY:
This is a prospective randomized, double-blind, placebo-controlled study in participants with disabling migraine (Migraine Disability Assessment (MIDAS) score ≥ 11).

DETAILED DESCRIPTION:
Participants will be asked to treat a migraine attack with study drug on an outpatient basis. Participants will be provided with a dosing card containing a dose for initial treatment and a second dose to be used for rescue or recurrence of migraine. Each participant's study participation will consist of screening (Visit 1) with a telephone contact within 7 days to confirm eligibility, a Treatment Period of up to 8 weeks, and End-of-Study (EoS) (Visit 2) within one week (7 days) of treating a single migraine attack. The total time on study is approximately up to 11 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent and authorize HIPAA.
* Participants with migraine with or without aura fulfilling the International Headache Society (IHS) diagnostic criteria 1.1 and 1.2.1 (International Headache Classification (ICHD) 2004).
* History of disabling migraine for at least 1 year.
* Migraine Disability Association (MIDAS) score ≥11.
* Migraine onset before the age of 50 years.
* History of 3 - 8 migraine attacks per month (< 15 headache days per month).
* Male or female, aged 18 years or above.
* Females of child-bearing potential must be using or willing to use a highly effective form of contraception (e.g. combined oral contraceptive, intrauterine device (IUD), abstinence or vasectomized partner).
* Able and willing to complete an electronic diary to record details of the migraine attack treated with study drug.

Exclusion Criteria:

* Any medical condition or clinical laboratory test which in the judgment of the Investigator makes the participant unsuitable for the study.
* Pregnant or breast-feeding women.
* Women of child-bearing potential not using or not willing to use highly effective contraception.
* Known hypersensitivity to lasmiditan or to any excipient of lasmiditan oral tablets, or any sensitivity to lasmiditan.
* History or evidence of hemorrhagic stroke, epilepsy or any other condition placing the participant at increased risk of seizures.
* History of recurrent dizziness and/or vertigo including benign paroxysmal positional vertigo (BPPV), Meniere's disease, vestibular migraine, and other vestibular disorders.
* History of diabetes mellitus with complications (diabetic retinopathy, nephropathy or neuropathy).
* History within the previous three years or current evidence of abuse of any drug, prescription or illicit, or alcohol.
* History of orthostatic hypotension with syncope.
* Significant renal or hepatic impairment.
* Participant is at imminent risk of suicide (positive response to question 4 or 5) on the Columbia-Suicide Severity Rating Scale (C-SSRS) or had a suicide attempt within six months prior to screening.
* Previous participation in this clinical trial.
* Participation in any clinical trial of an experimental drug or device in the previous 30 days.
* Known Hepatitis B or C or HIV infection.
* History, within past 12 months, of chronic migraine or other forms of primary or secondary chronic headache disorder (e.g. hemicranias continua, medication overuse headache) where headache frequency is ≥15 headache days per month.
* Use of more than 3 doses per month of either opiates or barbiturates.
* Initiation of or a change in concomitant medication to reduce the frequency of migraine episodes within three (3) months prior to Screening/Visit 1.
* Participants who are employees of the sponsor.
* Relatives of, or staff directly reporting to, the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3005 (Actual)
Dates: Start 2016-05; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (95):
- United States (95):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Medical Affiliated Research Center, Inc. - ARC, Huntsville, Alabama
  - 21st Century Neurology, Phoenix, Arizona
  - Anaheim Clinical Trials, Anaheim, California
  - The Research Center of Southern California, Carlsbad, California
  - eStudySite, Chula Vista, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, Newport Beach, California
  - Pacific Research Partners, Oakland, California
  - Desert Valley Research, Rancho Mirage, California
  - Northern California Clinical Research Center, Redding, California
  - Anderson Clinical Research, Redlands, California
  - California Research Foundation, San Diego, California
  - Neurological Research Institute, Santa Monica, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Encompass Clinical Research, Spring Valley, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Lytle and Weiss, PLLC dba Clinical Trials of the Rockies, Denver, Colorado
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Nova Clinical Reseach, LLC, Bradenton, Florida
  - PAB Clinical Research, Brandon, Florida
  - Meridien Research, Brooksville, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - The Core Research, Doral, Florida
  - Clinical Research West Coast, Fort Myers, Florida
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - Infinity Clinical Research, LLC, Hollywood, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Florida Clinical Research, Maitland, Florida
  - Pharmax Research Clinic, Inc., Miami, Florida
  - Prestige Clinical Research Center, Inc., Miami, Florida
  - Floriday Medical Center and Research, Inc., Miami, Florida
  - Veritas Research Corporation, Miami Lakes, Florida
  - Harmony Clinical Research Inc., North Miami Beach, Florida
  - Compass Research, LLC, Orlando, Florida
  - Clinical Research Center, LLC, Royal Palm Beach, Florida
  - Meridien Research, Inc., St. Petersburg, Florida
  - Meridian Clinical Research, LLC, Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Pinnacle Trials, Inc., Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Harbin Clinic, LLC, Rome, Georgia
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Meridian Clinical Research, Savannah, Georgia
  - Clinical Investigation Specialists, Inc., Gurnee, Illinois
  - Goldpoint Clinical Research, LLC, Indianapolis, Indiana
  - Heartland Research Associates, LLC, Augusta, Kansas
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Associates in Neurology, P.S.C., Lexington, Kentucky
  - Research Integrity, LLC., Owensboro, Kentucky
  - New Orleans Center for Clinical Research, Inc., New Orleans, Louisiana
  - Beacon Clinical Research, LLC, Quincy, Massachusetts
  - Michigan Head Pain & Neurological Institute, Ann Arbor, Michigan
  - Clinical Research Institute, Plymouth, Minnesota
  - Adirondack Medical Research Center, Omaha, Nebraska
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Regional Clinical Research, Inc., Endwell, New York
  - Rochester Clinical Research Inc., Rochester, New York
  - Asheville Neurology Specialists, PA, Asheville, North Carolina
  - PMG Research of Cary, LLC, Cary, North Carolina
  - Community Research, Cincinnati, Ohio
  - IVA Research, Cincinnati, Ohio
  - Summit Research Network (Oregon) Inc., Portland, Oregon
  - Partners in Clinical Research, Cumberland, Rhode Island
  - BTC of Lincoln Research,LLC, Lincoln, Rhode Island
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Mountain View Clinical Research, Inc., Greer, South Carolina
  - Coastal Carolina Research Center, Inc, Mt. Pleasant, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - ClinSearch, LLC, Chattanooga, Tennessee
  - Holston Medical Group, P.C., Kingsport, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Nashville Neuroscience Group, Nashville, Tennessee
  - Central Texas Clinical Research, LLC, Austin, Texas
  - FutureSearch Trials of Neurology, Austin, Texas
  - Tekton Research, Inc., Austin, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Protenium Clinical Research, Hurst, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Ericksen Research & Development, LLC, Clinton, Utah
  - J. Lewis Research, Inc. Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research Inc.- Foothill Family Clinic South, Salt Lake City, Utah
  - Jean Brown Research, Salt Lake City, Utah
  - Wasatch Clinical Research, Salt Lake City, Utah
  - J. Lewis Research, Inc. - Jordan River Family Medicine, South Jordan, Utah
  - Charlottesville Medical Research, LLC, Charlottesville, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - MultiCare Health System Institute for Research and Innovation, Tacoma, Washington
  - Clinical Investigation Specialists Inc, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Johnston KM, Powell L, Popoff E, Harris L, Croop R, Coric V, L'Italien G. Rimegepant, Ubrogepant, and Lasmiditan in the Acute Treatment of Migraine Examining the Benefit-Risk Profile Using Number Needed to Treat/Harm. Clin J Pain. 2022 Nov 1;38(11):680-685. doi: 10.1097/AJP.0000000000001072. PMID 36125279
- [Derived] Doty EG, Hauck PM, Krege JH, Komori M, Hake AM, Dong Y, Lipton RB. The Association Between the Occurrence of Common Treatment-Emergent Adverse Events and Efficacy Outcomes After Lasmiditan Treatment of a Single Migraine Attack: Secondary Analyses from Four Pooled Randomized Clinical Trials. CNS Drugs. 2022 Jul;36(7):771-783. doi: 10.1007/s40263-022-00928-y. Epub 2022 Jul 2. PMID 35779194
- [Derived] Krege JH, Lipton RB, Baygani SK, Komori M, Ryan SM, Vincent M. Lasmiditan for Patients with Migraine and Contraindications to Triptans: A Post Hoc Analysis. Pain Ther. 2022 Jun;11(2):701-712. doi: 10.1007/s40122-022-00388-8. Epub 2022 Apr 26. PMID 35471625
- [Derived] Charleston L 4th, Savage-Edwards B, Bragg SM, Baygani SK, Dennehy EB. Migraine history and response to lasmiditan across racial and ethnic groups. Curr Med Res Opin. 2022 May;38(5):721-730. doi: 10.1080/03007995.2022.2057152. Epub 2022 Apr 3. PMID 35350937
- [Derived] Reuter U, Krege JH, Lombard L, Gomez Valderas E, Krikke-Workel J, Dell-Agnello G, Dowsett SA, Buse DC. Lasmiditan efficacy in the acute treatment of migraine was independent of prior response to triptans: Findings from the CENTURION study. Cephalalgia. 2022 Jan;42(1):20-30. doi: 10.1177/03331024211048507. Epub 2021 Oct 13. PMID 34644189
- [Derived] Lipton RB, Baygani SK, Tepper SJ, Krege JH, Vasudeva R, Pearlman EM, Hauck PM, Loo LS. A close association of freedom from pain, migraine-related functional disability, and other outcomes: results of a post hoc analysis of randomized lasmiditan studies SAMURAI and SPARTAN. J Headache Pain. 2021 Aug 28;22(1):101. doi: 10.1186/s10194-021-01303-w. PMID 34454420
- [Derived] Martin VT, Ahmed Z, Hochstetler HM, Baygani SK, Dong Y, Hauck PM, Khanna R. Tolerability and Safety of Lasmiditan Treatment in Elderly Patients With Migraine: Post Hoc Analyses From Randomized Studies. Clin Ther. 2021 Jun;43(6):1066-1078. doi: 10.1016/j.clinthera.2021.04.004. Epub 2021 Aug 6. PMID 34366152
- [Derived] Peres MFP, Vasudeva R, Baygani SK, Dennehy EB, Vincent M, Friedman DI. Lasmiditan efficacy in migraine attacks with mild vs. moderate or severe pain. Curr Med Res Opin. 2021 Jun;37(6):1031-1038. doi: 10.1080/03007995.2021.1903846. Epub 2021 Apr 7. PMID 33784930
- [Derived] Clemow DB, Hochstetler HM, Dong Y, Hauck P, Peres MFP, Ailani J. Effect of a change in lasmiditan dose on efficacy and safety in patients with migraine. Postgrad Med. 2021 May;133(4):449-459. doi: 10.1080/00325481.2020.1860619. Epub 2021 Mar 17. PMID 33730977
- [Derived] Clemow DB, Baygani SK, Hauck PM, Hultman CB. Lasmiditan in patients with common migraine comorbidities: a post hoc efficacy and safety analysis of two phase 3 randomized clinical trials. Curr Med Res Opin. 2020 Nov;36(11):1791-1806. doi: 10.1080/03007995.2020.1808780. Epub 2020 Oct 6. PMID 32783644
- [Derived] Smith T, Krege JH, Rathmann SS, Dowsett SA, Hake A, Nery ESM, Matthews BR, Doty EG. Improvement in Function after Lasmiditan Treatment: Post Hoc Analysis of Data from Phase 3 Studies. Neurol Ther. 2020 Dec;9(2):459-471. doi: 10.1007/s40120-020-00185-5. Epub 2020 May 23. PMID 32447545
- [Derived] Knievel K, Buchanan AS, Lombard L, Baygani S, Raskin J, Krege JH, Loo LS, Komori M, Tobin J. Lasmiditan for the acute treatment of migraine: Subgroup analyses by prior response to triptans. Cephalalgia. 2020 Jan;40(1):19-27. doi: 10.1177/0333102419889350. Epub 2019 Nov 19. PMID 31744319
- [Derived] Ashina M, Vasudeva R, Jin L, Lombard L, Gray E, Doty EG, Yunes-Medina L, Kinchen KS, Tassorelli C. Onset of Efficacy Following Oral Treatment With Lasmiditan for the Acute Treatment of Migraine: Integrated Results From 2 Randomized Double-Blind Placebo-Controlled Phase 3 Clinical Studies. Headache. 2019 Nov;59(10):1788-1801. doi: 10.1111/head.13636. Epub 2019 Sep 17. PMID 31529622
- [Derived] Shapiro RE, Hochstetler HM, Dennehy EB, Khanna R, Doty EG, Berg PH, Starling AJ. Lasmiditan for acute treatment of migraine in patients with cardiovascular risk factors: post-hoc analysis of pooled results from 2 randomized, double-blind, placebo-controlled, phase 3 trials. J Headache Pain. 2019 Aug 29;20(1):90. doi: 10.1186/s10194-019-1044-6. PMID 31464581
- [Derived] Loo LS, Plato BM, Turner IM, Case MG, Raskin J, Dowsett SA, Krege JH. Effect of a rescue or recurrence dose of lasmiditan on efficacy and safety in the acute treatment of migraine: findings from the phase 3 trials (SAMURAI and SPARTAN). BMC Neurol. 2019 Aug 13;19(1):191. doi: 10.1186/s12883-019-1420-5. PMID 31409292
- [Derived] Loo LS, Ailani J, Schim J, Baygani S, Hundemer HP, Port M, Krege JH. Efficacy and safety of lasmiditan in patients using concomitant migraine preventive medications: findings from SAMURAI and SPARTAN, two randomized phase 3 trials. J Headache Pain. 2019 Jul 24;20(1):84. doi: 10.1186/s10194-019-1032-x. PMID 31340760
- [Derived] Doty EG, Krege JH, Jin L, Raskin J, Halker Singh RB, Kalidas K. Sustained responses to lasmiditan: Results from post-hoc analyses of two Phase 3 randomized clinical trials for acute treatment of migraine. Cephalalgia. 2019 Oct;39(12):1569-1576. doi: 10.1177/0333102419859313. Epub 2019 Jul 3. PMID 31266353
- [Derived] Krege JH, Rizzoli PB, Liffick E, Doty EG, Dowsett SA, Wang J, Buchanan AS. Safety findings from Phase 3 lasmiditan studies for acute treatment of migraine: Results from SAMURAI and SPARTAN. Cephalalgia. 2019 Jul;39(8):957-966. doi: 10.1177/0333102419855080. Epub 2019 Jun 5. PMID 31166697
- [Derived] Tepper SJ, Krege JH, Lombard L, Asafu-Adjei JK, Dowsett SA, Raskin J, Buchanan AS, Friedman DI. Characterization of Dizziness After Lasmiditan Usage: Findings From the SAMURAI and SPARTAN Acute Migraine Treatment Randomized Trials. Headache. 2019 Jul;59(7):1052-1062. doi: 10.1111/head.13544. Epub 2019 Jun 1. PMID 31152441

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomly assigned to 1 of 7 sequences and received lasmiditan 50 mg (L50 mg), lasmiditan 100 mg (L100 mg) or lasmiditan 200 mg (L200 mg) or placebo (P) for the first dose and the second dose, if needed for rescue or recurrence of migraine.
Groups:
- Lasmiditan 50 Milligram (mg)/Lasmiditan 50 mg: Lasmiditan 50 mg was administered orally, once for acute treatment of migraine. An optional second dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
- Lasmiditan 50 mg/Placebo: Lasmiditan 50 mg was administered orally, once for acute treatment of migraine. An optional placebo second dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
- Lasmiditan 100 mg/Lasmiditan 100 mg: Lasmiditan 100 mg was administered orally, once for acute treatment of migraine. An optional second dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
- Lasmitidan 100 mg/Placebo: Lasmiditan 100 mg was administered orally, once for acute treatment of migraine. An optional placebo second dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
- Lasmiditan 200 mg/Lasmiditan 200 mg: Lasmiditan 200 mg was administered orally, once for acute treatment of migraine. An optional second dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
- Lasmitidan 200 mg/Placebo: Lasmiditan 200 mg was administered orally, once for acute treatment of migraine. An optional placebo second dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
- Placebo/Placebo: Placebo tablets match each of the lasmiditan doses (50 mg, 100 mg and 200 mg) was administered orally, daily for acute treatment of migraine. An optional second dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
Period: Overall Study
Arm/Group | Lasmiditan 50 Milligram (mg)/Lasmiditan 50 mg | Lasmiditan 50 mg/Placebo | Lasmiditan 100 mg/Lasmiditan 100 mg | Lasmitidan 100 mg/Placebo | Lasmiditan 200 mg/Lasmiditan 200 mg | Lasmitidan 200 mg/Placebo | Placebo/Placebo
Started | 501 | 249 | 502 | 252 | 501 | 249 | 751
Received at Least 1 Dose of Study Drug | 429 | 225 | 423 | 212 | 434 | 215 | 645
Received Optional 2nd Dose | 206 | 96 | 177 | 83 | 144 | 74 | 361
Completed (One site was burned down and several participants have incomplete data.) | 437 | 226 | 426 | 216 | 448 | 217 | 662
Not Completed | 64 | 23 | 76 | 36 | 53 | 32 | 89
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 4 | 0 | 0
Not completed — Lost to Follow-up | 20 | 7 | 27 | 10 | 20 | 10 | 29
Not completed — Protocol Violation | 10 | 4 | 14 | 6 | 7 | 7 | 12
Not completed — Pregnancy | 1 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 6 | 14 | 11 | 6 | 4 | 15
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Randomization Failure | 22 | 6 | 20 | 7 | 16 | 11 | 30

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Lasmiditan 50 mg: Lasmiditan 50 mg was administered orally, once for acute treatment of migraine. A second optional dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
- Lasmiditan 100 mg: Lasmiditan 100 mg was administered orally, once for acute treatment of migraine. A second optional dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
- Lasmiditan 200 mg: Lasmiditan 200 mg was administered orally, once for acute treatment of migraine. A second optional dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
- Placebo: Placebo tablets match each of the lasmiditan doses (50 mg, 100 mg and 200 mg) was administered orally, once for acute treatment of migraine. A second optional dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
- Total: Total of all reporting groups
Arm/Group | Lasmiditan 50 mg | Lasmiditan 100 mg | Lasmiditan 200 mg | Placebo | Total
Number analyzed (Participants) | 654 | 635 | 649 | 645 | 2583
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (13.20) | 43.4 (12.59) | 41.8 (12.40) | 42.6 (12.90) | 42.7 (12.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 554 | 539 | 536 | 545 | 2174
  Male | 100 | 96 | 113 | 100 | 409
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 2 | 5 | 12
  Asian | 5 | 6 | 7 | 3 | 21
  Black or African American | 106 | 104 | 106 | 110 | 426
  Native Hawaiian or other Pacific Islander | 2 | 1 | 2 | 2 | 7
  White | 524 | 509 | 522 | 516 | 2071
  Other | 6 | 8 | 4 | 4 | 22
  Multiple | 8 | 5 | 5 | 5 | 23
  Missing | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 135 | 137 | 136 | 124 | 532
  Not Hispanic or Latino | 515 | 493 | 511 | 518 | 2037
  Not Reported | 3 | 3 | 0 | 3 | 9
  Unknown | 1 | 2 | 1 | 0 | 4
  Missing | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants] — Population: Participants in each region are those who were randomized to each arm.
  Participants
    Germany | 77 | 79 | 77 | 77 | 310
    United Kingdom | 48 | 48 | 47 | 48 | 191
    United States | 625 | 627 | 626 | 626 | 2504

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Headache Pain Free at 2 Hours Post Dose
Description: The percentage of participants defined as mild, moderate, or severe headache pain becoming none.
Time Frame: 2 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable headache pain free data.
Measure: Number; unit: percentage of participants
Groups:
- Lasmiditan 50 mg: Lasmiditan 50 mg was administered orally, once for acute treatment of migraine. A second dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
- Lasmiditan 100 mg: Lasmiditan 100 mg was administered orally, once for acute treatment of migraine. A second dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
- Lasmiditan 200 mg: Lasmiditan 200 mg was administered orally, once for acute treatment of migraine. A second dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
- Placebo: Placebo tablets match each of the lasmiditan doses (50 mg, 100 mg and 200 mg) was administered orally, once for acute treatment of migraine. A second dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
Arm/Group | Lasmiditan 50 mg | Lasmiditan 100 mg | Lasmiditan 200 mg | Placebo
Number analyzed (Participants) | 556 | 532 | 528 | 539
percentage of participants | 28.6 | 31.4 | 38.8 | 21.3
Statistical Analysis 1: Comparison: Lasmiditan 50 mg vs Placebo; Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 1.5, 95% CI 2-sided [1.1 to 1.9]
Statistical Analysis 2: Comparison: Lasmiditan 100 mg vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.7, 95% CI 2-sided [1.3 to 2.2]
Statistical Analysis 3: Comparison: Lasmiditan 200 mg vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.3, 95% CI 2-sided [1.8 to 3.1]

2. Primary Outcome: Percentage of Participants Who Are Most Bothersome Symptom (MBS) Free
Description: The percentage of participants defined as the associated symptom present and identified as MBS (nausea, photophobia, or phonophobia) prior to dosing being absent.
Time Frame: 2 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable MBS data.
Measure: Number; unit: percentage of participants
Arm/Group | Lasmiditan 50 mg | Lasmiditan 100 mg | Lasmiditan 200 mg | Placebo
Number analyzed (Participants) | 512 | 500 | 483 | 514
percentage of participants | 40.8 | 44.2 | 48.7 | 33.5
Statistical Analysis 1: Comparison: Lasmiditan 50 mg vs Placebo; Test type: Superiority; p = 0.009, Regression, Logistic; Odds Ratio (OR) = 1.4, 95% CI 2-sided [1.1 to 1.8]
Statistical Analysis 2: Comparison: Lasmiditan 100 mg vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.6, 95% CI 2-sided [1.2 to 2.0]
Statistical Analysis 3: Comparison: Lasmiditan 200 mg vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.9, 95% CI 2-sided [1.4 to 2.4]

3. Other Pre Specified Outcome: Percentage of Participants With Headache Relief
Description: The percentage of participants with headache pain moderate or severe which became mild or none or with headache pain mild which became none.
Time Frame: 2 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable headache relief data.
Measure: Number; unit: percentage of participants
Arm/Group | Lasmiditan 50 mg | Lasmiditan 100 mg | Lasmiditan 200 mg | Placebo
Number analyzed (Participants) | 598 | 571 | 565 | 575
percentage of participants | 59.0 | 64.8 | 65.0 | 47.7
Statistical Analysis 1: Comparison: Lasmiditan 50 mg vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.7, 95% CI 2-sided [1.3 to 2.2]
Statistical Analysis 2: Comparison: Lasmiditan 100 mg vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.3, 95% CI 2-sided [1.7 to 2.9]
Statistical Analysis 3: Comparison: Lasmiditan 200 mg vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.4, 95% CI 2-sided [1.8 to 3.1]

4. Other Pre Specified Outcome: Number of Participants With Headache Recurrence
Description: The number of participants with headache recurrence (moderate or severe at baseline which became pain-free at 2 hours post dose and worsened again up to 48 hours post dose)
Time Frame: From 2 Hours Post Dose Up to 48 Hours
Population: All randomized participants who received at least one dose of study drug and had evaluable headache recurrence data.
Measure: Count of Participants; unit: Participants
Arm/Group | Lasmiditan 50 mg | Lasmiditan 100 mg | Lasmiditan 200 mg | Placebo
Number analyzed (Participants) | 159 | 167 | 205 | 115
Participants | 38 | 44 | 52 | 26

5. Other Pre Specified Outcome: Percentage of Participants Use of Rescue Medication
Description: The percentage of participants who used rescue medication.
Time Frame: 2 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable use of rescue medication data.
Measure: Number; unit: percentage of participants
Arm/Group | Lasmiditan 50 mg | Lasmiditan 100 mg | Lasmiditan 200 mg | Placebo
Number analyzed (Participants) | 598 | 571 | 565 | 576
percentage of participants | 31.9 | 26.4 | 18.9 | 40.8
Statistical Analysis 1: Comparison: Lasmiditan 50 mg vs Placebo; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.5 to 0.9]
Statistical Analysis 2: Comparison: Lasmiditan 100 mg vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.5, 95% CI 2-sided [0.4 to 0.7]
Statistical Analysis 3: Comparison: Lasmiditan 200 mg vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.3, 95% CI 2-sided [0.3 to 0.4]

6. Other Pre Specified Outcome: Percentage of Participants Use of Rescue Medication
Description: The percentage of participants who used rescue medication.
Time Frame: From 2 Hours Post Dose Up to 24 Hours
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Lasmiditan 50 mg | Lasmiditan 100 mg | Lasmiditan 200 mg | Placebo
Number analyzed (Participants) | 598 | 571 | 565 | 576
percentage of participants | 8.9 | 6.3 | 7.4 | 8.7
Statistical Analysis 1: Comparison: Lasmiditan 50 mg vs Placebo; Test type: Superiority; p = 0.917, Regression, Logistic; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.7 to 1.5]
Statistical Analysis 2: Comparison: Lasmiditan 100 mg vs Placebo; Test type: Superiority; p = 0.129, Regression, Logistic; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.5 to 1.1]
Statistical Analysis 3: Comparison: Lasmiditan 200 mg vs Placebo; Test type: Superiority; p = 0.456, Regression, Logistic; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.6 to 1.3]

7. Other Pre Specified Outcome: Percentage of Participants Use of Rescue Medication
Description: The percentage of participants who used rescue medication.
Time Frame: From 24 Post Dose Up to 48 Hours
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Lasmiditan 50 mg | Lasmiditan 100 mg | Lasmiditan 200 mg | Placebo
Number analyzed (Participants) | 598 | 571 | 565 | 576
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

8. Other Pre Specified Outcome: Percentage of Participants Nausea Free
Description: The percentage of participant without nausea.
Time Frame: 2 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable nausea free data.
Measure: Number; unit: percentage of participants
Arm/Group | Lasmiditan 50 mg | Lasmiditan 100 mg | Lasmiditan 200 mg | Placebo
Number analyzed (Participants) | 598 | 571 | 565 | 576
percentage of participants | 68.7 | 71.8 | 70.4 | 70.3
Statistical Analysis 1: Comparison: Lasmiditan 50 mg vs Placebo; Test type: Superiority; p = 0.522, Regression, Logistic; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.7 to 1.2]
Statistical Analysis 2: Comparison: Lasmiditan 100 mg vs Placebo; Test type: Superiority; p = 0.622, Regression, Logistic; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.8 to 1.4]
Statistical Analysis 3: Comparison: Lasmiditan 200 mg vs Placebo; Test type: Superiority; p = 0.992, Regression, Logistic; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.8 to 1.3]

9. Other Pre Specified Outcome: Percentage of Participants With Phonophobia Free
Description: The percentage of participants without phonophobia.
Time Frame: 2 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable phonophobia free data.
Measure: Number; unit: percentage of participants
Arm/Group | Lasmiditan 50 mg | Lasmiditan 100 mg | Lasmiditan 200 mg | Placebo
Number analyzed (Participants) | 598 | 571 | 565 | 576
percentage of participants | 61.2 | 64.8 | 65.3 | 53.5
Statistical Analysis 1: Comparison: Lasmiditan 50 mg vs Placebo; Test type: Superiority; p = 0.008, Regression, Logistic; Odds Ratio (OR) = 1.4, 95% CI 2-sided [1.1 to 1.7]
Statistical Analysis 2: Comparison: Lasmiditan 100 mg vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.6, 95% CI 2-sided [1.3 to 2.0]
Statistical Analysis 3: Comparison: Lasmiditan 200 mg vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.6, 95% CI 2-sided [1.3 to 2.1]

10. Other Pre Specified Outcome: Percentage of Participants With Photophobia Free
Description: The percentage of participants without photophobia.
Time Frame: 2 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable photophobia free data.
Measure: Number; unit: percentage of participants
Arm/Group | Lasmiditan 50 mg | Lasmiditan 100 mg | Lasmiditan 200 mg | Placebo
Number analyzed (Participants) | 598 | 571 | 565 | 576
percentage of participants | 51.2 | 56.4 | 58.2 | 43.2
Statistical Analysis 1: Comparison: Lasmiditan 50 mg vs Placebo; Test type: Superiority; p = 0.007, Regression, Logistic; Odds Ratio (OR) = 1.4, 95% CI 2-sided [1.1 to 1.7]
Statistical Analysis 2: Comparison: Lasmiditan 100 mg vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.7, 95% CI 2-sided [1.3 to 2.1]
Statistical Analysis 3: Comparison: Lasmiditan 200 mg vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.8, 95% CI 2-sided [1.4 to 2.3]

11. Other Pre Specified Outcome: Percentage of Participants With Resource Utilization
Description: Use of health care for treatment 6 months prior to enrolling in the study and information reported during time on study
Time Frame: 6 Months Prior to Enrolling in Study to End of Study (Up to 11 Weeks) Within 7 Days of Treating a Single Migraine Attack
Population: All randomized participants who had received at least one dose of study drug and had evaluable resource utilization data.
Measure: Number; unit: percentage of participants
Groups:
- Lasmiditan 50 mg/Lasmiditan 50 mg: Lasmiditan 50 mg was administered orally, once for acute treatment of migraine. An optional Lasmitidan 50 mg second dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
- Lasmiditan 100 mg/Lasmiditan 100 mg: Lasmiditan 100 mg was administered orally, once for acute treatment of migraine. A second optional dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
- Lasmiditan 100 mg/Placebo: Lasmiditan 100 mg was administered orally, once for acute treatment of migraine. A second optional dose was administered between 2 and 24 hours for rescue or recurrence of migraine. Then, participants were assigned to placebo.
- Lasmiditan 200 mg/Lasmiditan 200 mg: Lasmiditan 200 mg was administered orally, once for acute treatment of migraine. A second optional dose was administered between 2 and 24 hours for rescue or recurrence of migraine. Then, participants were assigned to Lasmiditan 200 mg.
- Lasmiditan 200 mg/Placebo: Lasmiditan 200 mg was administered orally, once for acute treatment of migraine. A second optional dose was administered between 2 and 24 hours for rescue or recurrence of migraine. Then, participants were assigned to placebo.
- Placebo/Placebo: Placebo tablets match each of the lasmiditan doses (50 mg, 100 mg and 200 mg) was administered orally, once for acute treatment of migraine. A second optional dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
Arm/Group | Lasmiditan 50 mg/Lasmiditan 50 mg | Lasmiditan 50 mg/Placebo | Lasmiditan 100 mg/Lasmiditan 100 mg | Lasmiditan 100 mg/Placebo | Lasmiditan 200 mg/Lasmiditan 200 mg | Lasmiditan 200 mg/Placebo | Placebo/Placebo
Number analyzed (Participants) | 429 | 225 | 423 | 212 | 434 | 215 | 645
percentage of participants
  6 months prior to enrolling | 4.7 | 2.2 | 2.8 | 2.4 | 3.2 | 3.3 | 2.9
  During time of study | 0.5 | 0 | 0.5 | 0 | 0.9 | 0.5 | 0.6

12. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Events
Description: Safety and Tolerability was assessed by the number of participants with at least 1 treatment emergent event (TEAE). A summary of other non-serious adverse events and all serious adverse events, regardless of causality, is located in the Reported Adverse Events Section
Time Frame: From Baseline Up to End of Study (Up to 11 Weeks)
Population: All randomized participants who had received at least one dose of study drug. Results are displayed by the first dose taken.
Measure: Number; unit: participants
Groups:
- Lasmiditan 50 mg: Lasmiditan 50 mg was administered orally, once for acute treatment of migraine. An optional Lasmitidan 50 mg second dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
- Lasmiditan 100 mg: Lasmiditan 100 mg was administered orally, once for acute treatment of migraine. An optional placebo second dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
Arm/Group | Lasmiditan 50 mg | Lasmiditan 100 mg | Lasmiditan 200 mg | Placebo
Number analyzed (Participants) | 654 | 635 | 649 | 645
participants | 167 | 230 | 253 | 75

ADVERSE EVENTS:
Time Frame: From Baseline Up to End of Study (Up to 11 Weeks)
Description: The safety population includes all participants who received at least one dose of study drug and the optional second dose.
Groups:
- Lasmiditan 100 mg/Lasmiditan 100 mg: Lasmiditan 100 mg was administered orally, once for acute treatment of migraine. An optional Lasmitidan 100 mg second dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
- Lasmiditan 100 mg/Placebo: Lasmiditan 100 mg was administered orally, once for acute treatment of migraine. An optional placebo second dose was administered between 2 and 24 hours for rescue or recurrence of migraine
- Lasmiditan 200 mg/Lasmiditan 200 mg: Lasmiditan 200 mg was administered orally, once for acute treatment of migraine. An optional Lasmitidan 200 mg second dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
- Lasmiditan 200 mg/Placebo: Lasmiditan 200 mg was administered orally, once for acute treatment of migraine. An optional placebo second dose was administered between 2 and 24 hours for rescue or recurrence of migraine
- Placebo/Placebo: Placebo tablets match each of the lasmiditan doses (50 mg, 100 mg and 200 mg) was administered orally, once for acute treatment of migraine. A second optional dose was administered within 24 hours for rescue or recurrence of migraine.
Arm/Group | Lasmiditan 50 mg/Lasmiditan 50 mg | Lasmiditan 50 mg/Placebo | Lasmiditan 100 mg/Lasmiditan 100 mg | Lasmiditan 100 mg/Placebo | Lasmiditan 200 mg/Lasmiditan 200 mg | Lasmiditan 200 mg/Placebo | Placebo/Placebo
All-Cause Mortality (participants affected / at risk) | 0/429 | 0/225 | 0/423 | 0/212 | 0/435 | 0/217 | 0/646
Serious Adverse Events (participants affected / at risk) | 1/429 | 0/225 | 1/423 | 1/212 | 3/435 | 0/217 | 2/646
Other Adverse Events (participants affected / at risk) | 118/429 | 61/225 | 149/423 | 94/212 | 177/435 | 87/217 | 80/646
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lasmiditan 50 mg/Lasmiditan 50 mg (N=429) | Lasmiditan 50 mg/Placebo (N=225) | Lasmiditan 100 mg/Lasmiditan 100 mg (N=423) | Lasmiditan 100 mg/Placebo (N=212) | Lasmiditan 200 mg/Lasmiditan 200 mg (N=435) | Lasmiditan 200 mg/Placebo (N=217) | Placebo/Placebo (N=646)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somatisation disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lasmiditan 50 mg/Lasmiditan 50 mg (N=429) | Lasmiditan 50 mg/Placebo (N=225) | Lasmiditan 100 mg/Lasmiditan 100 mg (N=423) | Lasmiditan 100 mg/Placebo (N=212) | Lasmiditan 200 mg/Lasmiditan 200 mg (N=435) | Lasmiditan 200 mg/Placebo (N=217) | Placebo/Placebo (N=646)
Palpitations (Cardiac disorders) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (3) | 3 (3) | 2 (2) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chromatopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mydriasis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Strabismus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 12 (12) | 6 (6) | 13 (13) | 9 (9) | 14 (14) | 4 (4) | 9 (9)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 4 (4) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 3 (3)
Asthenia (General disorders) | 2 (2) | 2 (2) | 2 (2) | 4 (4) | 8 (8) | 4 (4) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 13 (13) | 7 (7) | 13 (13) | 15 (15) | 21 (21) | 12 (12) | 6 (6)
Feeling abnormal (General disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sense of oppression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pulse pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) | 4 (4) | 4 (4) | 7 (7) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aura (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Clumsiness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 39 (42) | 18 (19) | 77 (84) | 45 (45) | 89 (94) | 33 (33) | 16 (17)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Facial spasm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Formication (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Head discomfort (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 5 (6) | 5 (5) | 10 (10) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 7 (8) | 2 (2) | 4 (4) | 4 (4) | 7 (7) | 7 (7) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 11 (13) | 7 (7) | 21 (22) | 17 (17) | 30 (34) | 13 (14) | 6 (6)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sedation (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 24 (25) | 11 (11) | 21 (21) | 10 (10) | 34 (36) | 12 (12) | 13 (13)
Stupor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 2 (2) | 0 (0)
Vertigo cns origin (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adjustment disorder with anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 6 (6) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Burnout syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depersonalisation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Euphoric mood (Psychiatric disorders) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypervigilance (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Panic reaction (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep terror (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal odour (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3)
Hot flush (Vascular disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-11-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT02605174/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT02605174/SAP_001.pdf